CLINICAL TRIAL: NCT06324071
Title: A Double-blind Randomized Placebo-controlled Clinical Study to Verify the Efficacy of TetraSOD® in the Improvement of Semen Quality in Patients With iIdiopathic Infertility
Brief Title: Study to Verify the Efficacy of a Product Containing 125 mg of TetraSOD® for the Treatment of Male Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fitoplancton Marino, S.L. (Industry)
Collaborators: Fundacio Clinic Barcelona (Other); Fertypharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022_TSOD_125
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Male Infertility
Keywords: TetraSOD®; Idiopathic Male Infertility; Oxidative stress
MeSH Terms: conditions — Infertility, Male | interventions — salicylhydroxamic acid; Superoxide Dismutase; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Group supplemented with a daily dose of placebo
  Interventions: Dietary Supplement: Sham
- Experimental group (Experimental): Group supplemented with 125 mg/day of TetraSOD®
  Interventions: Dietary Supplement: Marine microalgae Tetraselmis chuii with high Superoxide Dismutase (SOD) activity

INTERVENTIONS:
Dietary Supplement: Sham — Participants in the Control group will receive a daily dose of placebo in a capsule during 90 days.
  Arms: Control group
Dietary Supplement: Marine microalgae Tetraselmis chuii with high Superoxide Dismutase (SOD) activity — Participants in the Experimental group will receive a daily dose of 125 mg of TetraSOD® in a capsule during 90 days.
  Other Names: TetraSOD®
  Arms: Experimental group

SUMMARY:
TetraSOD® is a unique marine phytoplankton (Tetraselmis chuii) SOD-rich ingredient that is grown under patent-protected technology exclusively designed by the company Fitoplancton Marino, S.L. (Spain). In a previous pilot trial, the ability of TetraSOD® (dose: 250 mg/day) to improve semen characteristics in idiopathic infertile men after three months of treatment was assessed, revealing significant improvements in almost all of the analyzed parameters. In a further clinical trial close to finish (ClinicalTrials.gov Identifier: NCT04864314) using the same dose, such positive results have been tested again in a higher number of patients, and additional parameters have been included in order to gain insights into the sperm physiological changes that underpin the improvement in semen quality. In this new clinical trial, an intermediate dose (125 mg/day) is going to be tested in an attempt to determine a range of TetraSOD® dosage being clinically active for the treatment of male infertility.

DETAILED DESCRIPTION:
Infertility is an increasing global public health problem present in about 15-20% of the population of reproductive age, affecting as many as 186 million people worldwide. A male factor is present in approximately 50% of the infertile couples, a large number of them of unknown or idiopathic origin.

Spermatogenesis is a complex biological process that requires a highly regulated genetic and hormonal program in a singular environment created by the interaction with different cell types to orchestrate a successful differentiation process. This process occurs periodically every 72 days during a man's fertile life. It has been demonstrated that semen quality is deteriorating over the time, perhaps as a result of exposure to several environmental factors related with lifestyle: drug use (such us tobacco, alcohol, marijuana, cocaine, opioids and anabolic agents), diet and overweight, disorders of the sleep-wake cycle and working conditions (continuous exposure to heat sources or toxic substances) that could impact both directly and indirectly on the complex process of spermatogenesis.

Currently, the impact of oxidative stress, a cellular state product of an imbalance between the generation of highly unstable molecules known as reactive oxygen species (ROS) and the antioxidant cellular capacity in male fertility is being deeply investigated. High levels of oxidative stress in semen have been associated with both lower sperm concentration, sperm motility and acrosome integrity and higher sperm DNA damage and mitochondrial activity. Recent clinical trials have demonstrated the high prevalence of sperm DNA damage by up to 80% of men diagnosed with idiopathic male infertility. This DNA damage produced during spermatogenesis or sperm maturation process could be the result of an increase of reactive oxygen species (ROS) in male reproductive tract, which are related to different known factors (chronic systemic disease, use of some drugs, radiation or pesticides, febrile processes, old age and environmental factors related to lifestyle: smoking, obesity, alcohol) and other unknown so far.

Antioxidant supplementation has gained relevance within routine practices in patients with reproductive problems. Different studies have shown the beneficial effect of antioxidant consumption against oxidative damage caused by environmental and pathological components, improving sperm characteristics associated with the seminal analysis. There are scientific evidences about the improvement of male fertility and higher rates of live newborn after antioxidant treatment in subfertile men.

TetraSOD® is a unique commercial product comprised of 100% lyophilized biomass of the marine microalgae Tetraselmis chuii strain CCFM03 (Culture Collection of Fitoplancton Marino 03), which is currently marketed for food and nutraceutical applications around the world by the company Fitoplancton Marino, S.L. This microalgae product is characterized by a high content in the antioxidant enzyme superoxide dismutase (SOD), as it is produced using own patent-protected technology developed by the company. Results of in vitro studies with human cell lines suggest that TetraSOD® stimulates the cellular protective mechanisms against oxidative stress. Moreover, results previously obtained in a pilot study with the highest dose of TetraSOD® (250 mg/day) were promising, since a high statistically significant response was observed in three of the four studied parameters after three months of treatment.

Taking into account these results, a new extended double-blind randomized and placebo-controlled clinical study has been performed to confirm the positive effects of dietary supplementation with 250 mg of TetraSOD® during 3 months (corresponding to the time of a complete spermatogenic cycle) in sperm quality.

The main objective of this new study is to check the usefulness of a lower dose of TetraSOD® (125 mg/day) in the improvement of sperm quality, including sperm DNA fragmentation. As previously mentioned, oxidative stress is one of the main causes of sperm DNA damage. Nowadays, a diagnostic test for the study of the sperm DNA fragmentation exists, but it requires a specific sperm sample processing and the results are obtained in delay-time. In this new trial, correlation between sperm DNA fragmentation and static oxidation reduction potential (sORP) degree by the use of the Male Infertility Oxidative System (MiOXSYS) will be also tested as in the previous one with a higher dose of TetraSOD® (250 mg/day). Classical seminal parameters (semen volume, sperm concentration and number, sperm progressive motility) will be also quantified. In that way, with this new trial it will be possible to determine a range of TetraSOD® dosage being clinically active for the treatment of male infertility.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45
* Male patients with idiopathic infertility classified with asthenozoospermia, oligozoospermia or oligoasthenozoospermia after seminal assessment.
* Not achieving pregnancy after at least one year of intercourse with the same partner without protective measures

Exclusion Criteria:

* Azoospermia (absence of spermatozoa) or severe oligozoospermia (< 5 x 10^6 spermatozoa/ml of ejaculate)
* Testicular torsion or prostatitis
* Urinary retention and infections
* Drug consumption
* Hormone treatments
* Recent surgical interventions
* Diabetes
* Kidney or liver disease
* Leukocytosis
* Antioxidant supplement consumption in the last 3 months
* BMI>30 Kg/m2
* Endocrinopathies, hypo and hyperthyroidism
* Chromosomal anomalies (XX, XYY, XXY)
* Treatments with anticoagulants
* Radiotherapy/Chemotherapy
* Participation in another clinical study prior to inclusion in this study that could affect the objectives of the current study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sperm motility | 90 days
  Sperm motility will be assessed according to the method described in the World Health Organization (WHO) laboratory manual for the examination and processing of human semen, 5th ed. Geneva: World Health Organization (2010)
Sperm concentration | 90 days
  Sperm concentration will be determined according to the method described in the WHO laboratory manual for the examination and processing of human semen, 5th ed. Geneva: World Health Organization (2010)
Sperm oxidative stress | 90 days
  Sperm ROS intracellular will be measured by flow cytometry evaluating the sperm intracellular ROS (superoxide anion, hydroxyl radical, hydrogen peroxide)

SECONDARY OUTCOMES:
DNA integrity | 90 days
  DNA integrity/fragmentation will be evaluated using the COMET assay
sORP by MiOXSYS | 90 days
  sORP will be also assessed using the MiOXSYS system
Adverse effects | 90 days
  Any kind of adverse event attributable to TetraSOD® will be recorded during the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Corral, Principal Investigator — Hospital Clinic Barcelona, Spain; Meritxell Jodar, Principal Investigator — Hospital Clinic Barcelona, Spain
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No